CLINICAL TRIAL: NCT00951067
Title: Trial to Compare Pneumatic Compression Treatments for Upper Extremity Acquired Lymphedema
Brief Title: Pneumatic Compression Treatment For Upper Extremity Acquired Lymphedema
Acronym: PCD-LYMPH
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding not available to continue with study.
Sponsor: Boston Children's Hospital (Other)
Collaborators: NormaTec Industries LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AQ-UE-LYMPHEDMA-PCD-RCT
Record Dates: First submitted 2009-08-03; First posted 2009-08-04 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2014-01

CONDITIONS: Lymphedema
Keywords: Lymphedema; Breast Cancer; Upper Extremity; Arm
MeSH Terms: conditions — Lymphedema; Breast Neoplasms | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group A (Active Comparator): Exercise, Elevation, and Garment Compression
  Interventions: Other: Exercise, Elevation, and Compression Garment
- Group B (Active Comparator): Pneumatic Compression Device (B)
  Interventions: Device: E0650 PCD with non-sequential waveform
- Group C (Active Comparator): Pneumatic Compression Device (C)
  Interventions: Device: E0651 PCD with sequential, non-gradient waveform
- Group D (Active Comparator): Pneumatic Compression Device (D)
  Interventions: Device: E0652 PCD with sequential, gradient waveform
- Group E (Active Comparator): Pneumatic Compression Device (E)
  Interventions: Device: E0652 PCD with peristaltic pulse waveform

INTERVENTIONS:
Other: Exercise, Elevation, and Compression Garment — Patients will be asked to daily:
  * exercise
  * elevate arm
  * wear an arm compression garment
  Arms: Group A
Device: E0650 PCD with non-sequential waveform — Use of an E0650 PCD with non-sequential waveform for two hours every day.
  Other Names: Brand: Huntleigh Flowtron Hydroven™ 3
  Arms: Group B
Device: E0651 PCD with sequential, non-gradient waveform — Use of an E0651 PCD with sequential, non-gradient waveform for two hours every day
  Other Names: Brand: Petite Basic System (Model 701A) Lympha Press
  Arms: Group C
Device: E0652 PCD with sequential, gradient waveform — Use of an E0652 PCD with sequential, gradient waveform for two hours every day.
  Other Names: Brand: Bio Compression Sequential Circulator 3008
  Arms: Group D
Device: E0652 PCD with peristaltic pulse waveform — Use the E0652 PCD with peristaltic pulse waveform for two hours every day.
  Other Names: NormaTec brand
  Arms: Group E

SUMMARY:
The purpose of this study is to determine how well different treatments for acquired lymphedema work.

The study will compare 5 different non-invasive treatments for acquired lymphedema of the arm to see which treats lymphedema best.

DETAILED DESCRIPTION:
This study will compare 5 non-invasive lymphedema treatments.

Patients will be assigned to either:

- A combination of arm exercises, arm elevation, and wearing of a compression garment every day

OR

- One of four possible pneumatic compression devices for just two hours every day.

Pneumatic compression devices are made up of an inflatable sleeve connected to a small controller unit that is plugged into the wall. They feel like having your blood pressure taken.

None of the treatments are experimental. None of the treatments are invasive. All the treatments are considered standard of care and are used in clinics throughout the United States. All of the treatments will be done at home.

The trial will last for 7 and 1/2 months and will require follow-up visits to monitor progress.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with acquired lymphedema of the arm.

Exclusion Criteria:

* Refusal of consent
* Unlikely compliance with the research protocol
* Acute upper extremity DVT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-08; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Arm Volume | Arm volume will be measured at 2 weeks before treatment starts, day treatment begins, and then 1 month, 3 months, 6 months, and 7 months after treatment starts

SECONDARY OUTCOMES:
Infection (cellulitis) | Presence of infection will be recorded at 2 weeks before treatment starts, day treatment begins, and then 1 month, 3 months, 6 months, and 7 months after treatment starts
Quality of Life Survey | Survey will be given at 2 weeks before treatment starts, day treatment begins, and then 1 month, 3 months, 6 months, and 7 months after treatment starts

CONTACTS AND LOCATIONS:
Overall Officials: Arin K Greene, MD, MMSc, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston at Waltham, Waltham, Massachusetts, United States